CLINICAL TRIAL: NCT00001317
Title: A Phase IV Study of Recombinant Human Gamma Interferon in Patients With Chronic Granulomatous Diseases of Childhood
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 920186; 92-I-0186
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2000-05

CONDITIONS: Chronic Granulomatous Disease
Keywords: Children; Gamma Interferon; Hospitalizations; Infection; Chronic Granulomatous Disease
MeSH Terms: conditions — Granulomatous Disease, Chronic; Infections | interventions — Interferon-gamma

INTERVENTIONS:
Drug: interferon-gamma

SUMMARY:
In a recent double-blinded, placebo-controlled multi-center international study, subcutaneous injections of interferon-gamma administered three times weekly reduced the frequency of serious infections in patients with chronic granulomatous disease. Patients receiving interferon-gamma had fewer hospital stays, shorter in length, than the placebo group. Children less than 10 years of age benefitted most from treatment and had fewer side effects.

Based on these data, the FDA licensed interferon-gamma for prophylaxis in CGD patients. We wish to monitor our patients who participated in the original study for possible long-term side effects. Any new patients referred to us who are either on interferon-gamma or considered to be candidates for interferon-gamma will be considered for this protocol. In addition, our patients who were originally accepted under Genentech's compassionate plea protocol will also be monitored under this new protocol. The patients will be evaluated every six months, with blood work and interim medical histories taken.

DETAILED DESCRIPTION:
In a recent double-blinded, placebo-controlled multi-center international study, subcutaneous injections of interferon-gamma administered three times weekly reduced the frequency of serious infections in patients with chronic granulomatous disease. Patients receiving interferon-gamma had fewer hospital stays, shorter in length, than the placebo group. Children less than 10 years of age benefitted most from treatment and had fewer side effects.

Based on these data, the FDA licensed interferon-gamma for prophylaxis in CGD patients. We wish to monitor our patients who participated in the original study for possible long-term side effects. Any new patients referred to us who are either on interferon-gamma or considered to be candidates for interferon-gamma will be considered for this protocol. In addition, our patients who were originally accepted under Genentech's compassionate plea protocol will also be monitored under this new protocol. The patients will be evaluated every six months, with blood work and interim medical histories taken.

ELIGIBILITY:
The diagnosis of chronic granulomatous disease as indicated by an unusual pattern of infection in the patient or one pedigree relation, confirmed by both of the following tests:

Abnormal neutrophil NBT slide test (following PMA stimulation) and neutrophil superoxide anion production less than or equal to 20 percent normal.

Preserved renal function (creatinine less than or equal to 2.0 mg/100 mL; less than or equal to 2+ proteinuria).

Preserved hepatic function (bilirubin less than or equal to 1.5 mg/100 mL; prothrombin time less than or equal to 1.3 x control).

Preserved hematologic function (WBC greater than or equal to 3000/mm3; granulocytes greater than 1500/mm3; platelets greater than or equal to 100,000/mm3).

A minimum life expectancy of three months.

Patients seropositive for Hepatitis B surface antigen may be entered but serum specimens for rIFN-y antibody should not be collected.

Patients must not be pregnant or lactating.

Patients of childbearing potential may be entered if using effective contraception.

Full recovery from previous serious infections requiring hospitalization and parenteral antibiotic therapy. At least two weeks must elapse following the cessation of parenteral antibiotic therapy before study admission.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 1992-05; Study Completion 2001-07

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Allergy and Infectious Diseases (NIAID), Bethesda, Maryland, United States

REFERENCES:
- [Background] Ross JP, Holland SM, Gill VJ, DeCarlo ES, Gallin JI. Severe Burkholderia (Pseudomonas) gladioli infection in chronic granulomatous disease: report of two successfully treated cases. Clin Infect Dis. 1995 Nov;21(5):1291-3. doi: 10.1093/clinids/21.5.1291. PMID 8589158
- [Background] Gallin JI, Farber JM, Holland SM, Nutman TB. Interferon-gamma in the management of infectious diseases. Ann Intern Med. 1995 Aug 1;123(3):216-24. doi: 10.7326/0003-4819-123-3-199508010-00009. PMID 7598304